CLINICAL TRIAL: NCT03992599
Title: Prospective Study of Oncologic Outcomes After Laparoscopic Modified Complete Mesocolic Excision for Non-metastatic Right Colon Cancer [PIONEER Study]: Multicenter, Single-Arm Study
Brief Title: Prospective Study of Oncologic Outcomes After Laparoscopic Modified Complete Mesocolic Excision for Non-metastatic Right Colon Cancer [PIONEER Study]
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2018-1162
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Adenocarcinoma of the Colon
Keywords: Adenocarcinoma in right colon; mCME; oncologic outcomes; right-sided colon cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Laparoscopic modified central mesocolic excision: Patients receiving laparoscopic colectomy with the concept of modified complete mesocolic excision for right-sided colon cancer
  Interventions: Procedure: Laparoscopic modified complete mesocolic excision

INTERVENTIONS:
Procedure: Laparoscopic modified complete mesocolic excision — First, complete kocherization may be required to clear possible tumor spread if the tumor is infiltrating or adhering to the duodenum or perinephric fat tissue. Second, if the tumor is locally advanced, the entire prerenal soft tissue behind Gerota's fascia may need to be cleared, especially for tumors growing toward the posterior. The third difference of mCME with the conventional CME involves the tailored resection of the mesocolon and ileal mesentery according to tumor location. After identifying the root of the middle colic artery, the site of the vascular ligation depends on the location of the tumor. When the tumor is located in the cecum and ascending colon, only the right branch of the middle colic artery is ligated. If the tumor was present in these latter sites, the root of the middle colic artery is ligated.
  Other Names: Laparoscopic right hemicolectomy

SUMMARY:
This study is a multi-institutional, prospective, observational study evaluation oncologic outcomes of laparoscopic modified complete mesocolic excision (mCME) on right-sided colon cancer.

The primary outcome of this study is 3 year disease-free survival. Secondary outcome measures include 3 year overall survival, incidence of surgical complications, completeness of mCME, and distribution of metastatic lymph nodes.

DETAILED DESCRIPTION:
The present study aims to evaluate the oncological outcomes of laparoscopic mCME on right-sided colon cancer. The right side of the colon was defined as the colon from cecum up to the proximal half of the transverse colon. The number of patients needs to get a 90% power is 250. Patients will be enrolled at five leading centers in South Korea. A complete information leaflet will give to the patients during the first consultation, which will correspond to the enrollment day. The preoperative, intraoperative, and postoperative period will be in complete accordance with the usual care of the center. The baseline demographics and conditions, as well as the perioperative items and the postoperative occurrences, will be recorded through a prior designed case report form. The follow-up encompasses 13 postoperative consultations: 1month, 3 months, after that every 3 months until 36 months.

The primary outcome of this study is 3-year disease-free survival. Secondary outcome measures include 3-year overall survival, the incidence of surgical complications, completeness of mCME, and distribution of metastatic lymph nodes. Review of resected surgical specimens and the operative field after completion of lymph node dissection will be done based on photographs to assess the quality if surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1. Qualitative diagnosis: a pathological diagnosis of adenocarcinoma; the tumor located between the cecum and the right 1/2 of transverse colon
* 2. Patients suitable for curative surgery older than 19 years old
* 3. ASA grade I-III
* 4. Patients without preoperative treatment
* 5. Informed consent

Exclusion Criteria:

* 1. Informed consent refusal
* 2. Patients who need emergency operation; such as perforation, malignant colonic obstruction
* 3. Preoperative imaging examination results show: distant metastasis
* 4. Hereditary colon cancer
* 5. History of any other malignant tumor in recent 5 years, except for cervical carcinoma in situ which has been cured, basal cell carcinoma or squamous cell carcinoma of skin;
* 6. Simultaneous or simultaneous multiple primary colorectal cancer
* 7. Women during Pregnancy or breast feeding period

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with adenocarcinoma arising from the right side of the colon who received laparoscopic mCME. The right side of the colon was defined as the colon from cecum up to the proximal half of transverse colon
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
3 year disease-free survival (DFS) | DFS will be measured up to three years after surgery, and the last visit is 14th visit after index surgery.
  The 3 year disease-free survival is defined as the time from surgery until documented recurrence or death from any cause.

SECONDARY OUTCOMES:
3 year overall survival (OS) | Three years after surgery
  The time from surgery until documented death from any cause
Incidence of surgical complications | Until four weeks after surgery
Completeness of mCME | Two weeks after surgery
  A. By reviewing resected surgical specimens based on photographs B. By reviewing the operative field after lymph node dissection and specimen removal based on photographs
Distribution of metastatic LNs | Two weeks after surgery
  Lymph nodes retrieved from resected surgical specimens to categorise

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Colon and Rectal Surgery, Department of Surgery, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang SY, Kim MJ, Kye BH, Han YD, Cho MS, Jeong SY, Cho HM, Kim H, Kang GH, Song SH, Park JS, Kim JS, Park SY, Kim J, Min BS. Prospective study of oncologic outcomes after laparoscopic modified complete mesocolic excision for non-metastatic right colon cancer (PIONEER study): study protocol of a multicentre single-arm trial. BMC Cancer. 2020 Jul 14;20(1):657. doi: 10.1186/s12885-020-07151-2. PMID 32664881